CLINICAL TRIAL: NCT06210594
Title: SHIELD (Staph Intervention for Effective Local Defense): An Open-label Randomized Controlled Trial to Assess Efficacy of a Sustained Intervention (Topical Antibiotics and Skin Antisepsis) to Decrease Staphylococcus Aureus Carriage in Adults
Brief Title: Staph Intervention for Effective Local Defense
Acronym: SHIELD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00027090; 5S06GM142120 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Skin and soft tissue infections (SSTI); Methicillin-resistant staphylococcus aureus (MRSA); Carriage density; Biomedical intervention
MeSH Terms: conditions — Staphylococcal Infections; Soft Tissue Infections | interventions — Mupirocin; chlorhexidine gluconate; Educational Status; Household Products

STUDY DESIGN:
Intervention Model Description: This study will be an open-label randomized controlled trial to determine the feasibility, acceptability, and efficacy of a carriage suppression regimen in reducing the prevalence of SA carriage and SA infections among adults at high risk of SA infections who are currently carrying SA in the oropharynx or anterior nares. Participants will be randomized in a ratio of 1:1 to either:
  1. education about SA and receipt of household supplies to reduce SA transmission in the home plus use of a nasal antibiotic twice daily for 5 days then maintenance with an antiseptic regimen (N=50; intervention group);
     or
  2. education/household supplies alone (N = 50; control group).
  All participants will be followed for 4 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education + Household supplies + Nasal antibiotic + Antiseptic regimen (Experimental): Participants in this arm will receive education about SA and household supplies (e.g., cleaning products, pump lotion, laundry detergent, towels) plus use of a nasal antibiotic (mupirocin) twice daily for 5 days then maintenance with an antiseptic regimen (Nozin twice daily plus chlorhexidine gluconate wash 3 times per week)
  Interventions: Combination Product: Mupirocin + Nozin + chlorhexidine gluconate; Behavioral: Education + Household supplies
- Education + Household supplies (Active Comparator): Participants in this arm will receive education about SA and household supplies (e.g., cleaning products, pump lotion, laundry detergent, towels).
  Interventions: Behavioral: Education + Household supplies

INTERVENTIONS:
Combination Product: Mupirocin + Nozin + chlorhexidine gluconate — Education/household supplies + antibiotic + antiseptic regimen
  Other Names: Bactroban + Nozin + Hibiclens
  Arms: Education + Household supplies + Nasal antibiotic + Antiseptic regimen
Behavioral: Education + Household supplies — Education/household supplies

SUMMARY:
Indigenous persons experience a high burden of Staphylococcus aureus (SA) invasive disease and skin and soft tissue infections. SA carriage on the skin is factor for development of SA infections. The goal of this clinical trial is to evaluate a community-informed approach to reduce carriage of SA. Participants will be assigned to education and household supplies for prevention of SA with and without a biomedical intervention. Researchers will compare SA carriage in the two groups.

DETAILED DESCRIPTION:
Staphylococcus aureus (SA) is a common cause of skin and soft tissue infections (SSTI) and invasive infections in the United States (US). Infections caused by methicillin-resistant SA (MRSA) are of particular concern because MRSA is harder to treat and associated with significant costs to healthcare systems and patients. The White Mountain Apache (WMA) Tribe experiences a higher burden of SA and MRSA infections than the general US population. Most cases of invasive SA occurred among adults with underlying conditions and led to significant morbidity.

SA carriage is an important factor for development of SA infections. When individuals or the household contacts have recurrent SA infections, the use of antimicrobial or antiseptic agents to suppress or eliminate SA carriage (so called "decolonization") may be recommended to help prevent infection. While there are several regimens available to suppress carriage, each has limitations (e.g., potential antimicrobial resistance following repeated use of mupirocin antibiotic ointment, lack of access to a bathtub or reliable water supply for bleach baths). These interventions are typically used over a short period of time (e.g., one-time administration over 5-10 days). Re-acquisition of carriage in the months following completion of the carriage suppression regimen is common. Use of the standard approaches to SA carriage suppression in the WMA community has been inconsistent and has been insufficient to control SA disease. New approaches are urgently needed.

In formative research conducted by the study team, in-depth interviews and focus group discussions were conducted with healthcare providers and community members to understand the culture and context of tribal communities as related to SA infections, disease, and prevention. The researchers found that there are gaps in community knowledge about SA as a cause of skin infections and how to prevent an infection. When asked about preferred method of intervention to reduce SA carriage, participants indicated a preference for the antiseptic nasal spray (daily use) and antiseptic body wash (regular use), which were easily administered and could be incorporated into a daily routine.

In this study, the investigators will conduct an open-label randomized controlled trial to determine the feasibility, acceptability, and efficacy of a carriage suppression regimen in reducing the prevalence of SA carriage and SA infections among adults at high risk of SA infections who are currently carrying SA on the skin. Following informed consent, participants will be randomized in a ratio of 1:1 to either: A) education about SA and receipt of household supplies to reduce SA transmission in the home plus use of a nasal antibiotic twice daily for 5 days then maintenance with an antiseptic regimen (N = 50; Group A); or B) education/household supplies alone (N = 50; Group B). The antiseptic regimen will consist of twice daily Nozin nasal antiseptic plus chlorhexidine gluconate wash three times a week. Participants assigned to Group A will continue the antiseptic regimen for 4 months. All participants will be followed for 4 months.

Study visits will occur at baseline (Day 0) and Days 14, 30, 60, 90, and 120. At each visit, a questionnaire will be administered and swabs will be collected at common carriage sites on the body (anterior nares, oropharynx, and groin). Group A will also receive reminder text messages or phone calls at a frequency of choice (e.g., once per day or once per week). After the Day 0 and Day 120 visits, the participant's medical record will be reviewed to document relevant medical history and outpatient and inpatient visits for SSTI and SA-related infections.

A home visit will be scheduled after Day 0 to collect environmental swabs at frequent hand-contact sites (e.g., bedroom, living room, bathroom) and swabs from indoor pet cats and dogs (e.g., dorsal fur and skin of groin). Household members will also be recruited to complete a brief questionnaire and sample collection (anterior nares, oropharynx, and groin).

A qualitative assessment will be conducted in a subset of index participants (n=6-10) in Group A to assess adherence and acceptability of the prevention regimen. Participants will be chosen using purposive sampling to represent a range of reported adherence at the D60 visit and invited to provide informed consent. The qualitative assessment will consist of one in-depth interview at the endpoint (4 months).

ELIGIBILITY:
Inclusion Criteria:

* Native American adult living on or adjacent to the WMA Tribal lands
* 18 years of age and older
* Lab-confirmed SA carriage at time of enrollment
* Ability to provide written informed consent
* Ability to comply with follow-up activities
* Risk factor for SA-associated infection: Diagnosed with diabetes OR body mass index ≥30 OR documented SSTI or SA infection in the past 3 years

Exclusion Criteria:

* Immediate family member of study staff
* Allergy to citrus or any ingredient in Nozin, Hibiclens, or mupirocin
* Without a permanent home (e.g., living in a group home, shelter, or is unhoused)
* Use of antibiotics within 30 days prior to the first study visit (time-limited)
* Current SA infection (time-limited)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of SA carriage | 4 months after randomization
  Compare SA carriage prevalence in the nose, throat, and skin (any site) between arms.

SECONDARY OUTCOMES:
Feasibility and Acceptability | 4 months
  Proportion adhering to intervention.
Feasibility and Acceptability as assessed by in depth interviews | 4 months
  Assess the feasibility and acceptability qualitatively through in-depth interviews (with a subset of participants).
Incidence of SSTI | 4 months
  Compare the incidence of skin and soft tissue infections (all cause) between arms.
Characterize SA isolates | 4 months
  Characterize SA isolates, including lineages (proportion belonging to each clonal complex) and antimicrobial resistance (proportion MRSA), during follow-up in both arms.
Confirmed SA infection | 4 months
  Compare the incidence of lab-confirmed SA infection (all types and SSTI separately) between arms.
Prevalence of SA carriage in index participants, household members, indoor pets, and household surfaces | Baseline, day 14, day 30, day 60, day 90, day 120
  Describe baseline prevalence of SA carriage in index patients, household members, indoor pets, and household surfaces, and longitudinal prevalence in index participants, and compare between arms.
Adverse events | 4 months
  The proportion of participants with adverse events (e.g., dry skin) and compare between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Hammitt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Whiteriver Center for Indigenous Health, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No